CLINICAL TRIAL: NCT00224731
Title: Sleep Disorders in Children With ADHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvolby, Allan, M.D. (Individual)
Other Study IDs: M-2549-03
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2005-09

CONDITIONS: Attention Disorder With Hyperactivity (ADHD)
Keywords: Attention disorder with hyperactivity; sleep; stimulants; actigraphy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
ADHD is often associated with sleep difficulties. Attention-deficit/hyperactivity disorder (ADHD) is the most common problem presented to children mental health services. The disorder affects approximately 5 % of school-age children. The core symptoms of this disorder include varying degrees of inattention, impulsiveness and restlessness.

In addition to the core symptoms, ADHD is associated with other problems (e.g. academic underachievement, poor social relations and sleep disturbances).

Despite clinical observations of sleep problems in children with ADHD, there is little empirical research on this topic. The prevalence, type of sleep problems, and significance of these sleep disturbances in children with ADHD remain undocumented.

The objective is to determine the relationship of sleep problems to attention deficit/hyperactive disorder, comorbid disorders, and the effect of stimulant treatment.

ELIGIBILITY:
Inclusion Criteria:

- We will compare a group of children with ADHD, other psychiatric disorder, and a healthy group of children age 5 - 10

Exclusion Criteria:

mental retardation -

Ages: 5 Years to 10 Years | Sex: All
Age Groups: Child
Enrollment: 100
Dates: Start 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: allan hvolby, M.D, Principal Investigator — child psychiatric department, Esbjerg
Locations (1):
- Child psychiatric department and University of southern Denmark, Esbjerg, Denmark

REFERENCES:
- [Derived] Hvolby A, Jorgensen J, Bilenberg N. Actigraphic and parental reports of sleep difficulties in children with attention-deficit/hyperactivity disorder. Arch Pediatr Adolesc Med. 2008 Apr;162(4):323-9. doi: 10.1001/archpedi.162.4.323. PMID 18391140